CLINICAL TRIAL: NCT05796271
Title: Clinical Trial of Roflumilast Added to Standard Chemoimmunotherapy for High-risk Diffuse Large B-cell Lymphoma (CTMS# 22-0016)
Brief Title: Clinical Trial of Roflumilast Added to Standard Chemoimmunotherapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate funding to begin enrolling subjects
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 22-0016
Record Dates: First submitted 2023-02-09; First posted 2023-04-03 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- R-Chop and Roflumilast (Experimental): All subjects will receive R-CHOP therapy at standard doses according to the standard preparation and infusion procedures of each investigational site, which is to be repeated every 21 days (+/- 3 days) for a total of 6 cycles. All subjects will receive a fixed oral dose of one 500 microgram (μg) tablet of roflumilast per day with or without food for all 21 days of each cycle, which will amount to a total of 126 doses. Subjects will be asked to keep a drug diary to record the days and times when Roflumilast is taken. The first dose will be given on the day of the first R-CHOP treatment.
  Interventions: Drug: R-Chop and Roflumilast

INTERVENTIONS:
Drug: R-Chop and Roflumilast — All subjects will receive R-CHOP therapy at standard doses according to the standard preparation and infusion procedures of each investigational site, which is to be repeated every 21 days (+/- 3 days) for a total of 6 cycles. All subjects will receive a fixed oral dose of one 500 microgram (μg) tablet of roflumilast per day with or without food for all 21 days of each cycle, which will amount to a total of 126 doses. Subjects will be asked to keep a drug diary to record the days and times when Roflumilast is taken. The first dose will be given on the day of the first R-CHOP treatment.
  Other Names: Daliresp

SUMMARY:
This study is an investigator-initiated, phase II, single arm, open label clinical trial that will enroll subjects with untreated diffuse large B-cell lymphoma (DLCBL) at moderate or high risk for poor outcome, defined as an NCCN-IPI score of 2 or higher. All subjects will receive investigational drug, and outcomes will be compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years of age or older.
2. Pathologically proven diffuse large B-cell lymphoma.
3. No prior systemic therapy for lymphoma.
4. Patient has provided informed consent.
5. Patient is willing and able to comply with clinic visits and procedure outlined in the study protocol.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Life expectancy of ≥3 months.
8. Ann Arbor stage II-IV
9. NCCN-IPI risk score of ≥ 2
10. Measurable disease, meaning at least 1 lymph node or other lymphomatous lesion with a long axis of ≥1.5 cm by CT imaging, and at least one FDG-avid lesion by FDG-PET scan.
11. Left ventricular ejection fraction of at least 45% by either echocardiography or radionucleotide angiography.
12. Ability to swallow oral tablets without difficulty.
13. All subjects with preserved reproductive potential must agree to practice abstinence or employ contraceptive measures for the duration of treatment and for 4 weeks following final dosing. All male subjects are considered to have reproductive potential. Female subjects of reproductive potential are those who: 1) are not at least 50 years old and have no menses for 24 consecutive months; or 2) have not been rendered surgically sterile (having undergone hysterectomy and/or bilateral salpingo-oophorectomy). Female subjects of reproductive potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (hCG) within 7 days of first day of drug dosing.
14. Meet the following clinical laboratory requirements:

    * Creatinine clearance ≥30 ml/min by Cockcroft-Gault formula;
    * Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (unless indirect bilirubin is elevated due to Gilbert's syndrome or hemolysis);
    * AST and ALT≤ 3 × ULN;
    * Platelet count ≥ 50,000/μL, with or without transfusion support;
    * ANC ≥ 1000/μL, with or without chronic granulocyte growth factor support;
    * Hemoglobin ≥8 g/dL, with or without transfusion support.

Exclusion Criteria:

2. Any active malignancy other than DLBCL 3. High grade B Cell Lymphoma with rearrangements of MYC and BCL2, MYC and BCL6, and /or MYC and BCL2/BCL6 ("double-hit" or "triple-hit" DLBCL) 4. Current participation in another interventional clinical study 5. Prior allogeneic bone marrow transplant within 12 months of screening date. 6. Prior autologous stem cell transplant within 6 months of screening date. 7. Immunotherapy, chemotherapy, radiotherapy, or investigational therapy within 6 months prior to drug dosing.

8. Active central nervous system (CNS) involvement by lymphoma, including untreated symptomatic epidural disease 9. Active uncontrolled infection. 10. Poorly controlled depressive symptoms and/or currently under management for depression that is poorly controlled.

11. Significant disease or medical conditions, as assessed by the Investigator and Sponsor, that would substantially increase the risk-benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, and congestive heart failure New York Heart Association Class III-IV.

12. Second malignancy, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancies for which subjects are not on active anti-cancer therapies and have had no evidence of active malignancy for at least 1 year.

13. History of major surgery within 3 weeks or minor surgery within 1 week of roflumilast administration. Major surgery includes, for example, any open or laparoscopic entry into a body cavity, or operative repair of fracture; minor surgery includes, for example, open surgical biopsy of palpable/superficial lymph node, or placement of vascular access device.

14. Other medical or psychiatric illness or organ dysfunction, which in the opinion of the investigator, would either compromise the subject's safety or interfere with the evaluation of the safety of the study agent.

15. Corrected QT interval (QTc) prolongation (defined as a QTc >450 ms for males and >470 ms for females Fridericia's correction) or other clinically significant ECG abnormalities as assessed by the investigator.

16. Baseline serum troponin above the upper limit of normal. 17. Baseline serum BNP above the age-adjusted upper limit of normal. 18. Baseline amylase above the upper limit of normal. 19. Subjects known to be HIV-positive must not have multi-drug resistant HIV infection, CD4 counts < 150/μl or other concurrent AIDS-defining conditions. Serologic screening for HIV is required within the 6 months prior to study enrollment.

20. Subjects positive for Hepatitis B surface antigen (HBsAg) or Hepatitis C-virus ribonucleic acid (HCV RNA), unless both AST and ALT≤1.25 x ULN and there is no known history of chronic active hepatitis. Serologic screening for hepatitis B and C testing is required within the 6 months prior to study enrollment.

21. Subjects with moderate or severe liver impairment, as defined by a Child-Pugh class of B or C.

22. Women who are pregnant or breastfeeding. 23. Current use of any of the following medications: boceprevir, carbamazepine, ciprofloxacin, cobicistat, conivaptan, enzalutamide, fluvoxamine, itraconazole, ketoconazole, mitotane, phenytoin, posaconazole, rifampin, ritonavir, St. John's Wort, telaprevir, voriconazole, or zafirlukast.

24. Current use of non-nucleoside reverse transcriptase inhibitors (NNRTI) including efavirenz, rilpivirine, etravirine, delavirdine, nevirapine, and lersivirine.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Anti-tumor efficacy: progression-free survival (PFS) | Measured every 3 weeks for 21 day cycles for the duration of study treatment, from Baseline to approximately one year
  To assess the change in anti-tumor efficacy of Roflumilast in combination with R-CHOP in subjects with previously untreated high-risk DLBCL who are appropriate for treatment by estimates of progression-free survival (PFS).

CONTACTS AND LOCATIONS:
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in publication will be shared at the end of the study.
Supporting Information: Study Protocol, SAP
Time Frame: At study end upon approval for publication